CLINICAL TRIAL: NCT02535884
Title: Deep Brain Stimulation (DBS) of the Globus Pallidus (GP) in Huntington's Disease (HD): A Prospective, Randomised, Controlled, International, Multi-centre Study
Brief Title: Deep Brain Stimulation (DBS) of the Globus Pallidus (GP) in Huntington's Disease (HD)
Acronym: HD-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: KKS Netzwerk (Network); Medtronic (Industry); The George Institute (Other); Egyptian Society of Neurological Surgeons (Other); CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KKS-198; DRKS00006785 (Registry Identifier: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; DBS; Chorea
MeSH Terms: conditions — Huntington Disease; Chorea

STUDY DESIGN:
Intervention Model Description: During the first 3 month the one group will be stimulated (pallidal DBS), thereafter 12 weeks open follow up, where patients in both groups are stimulated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stimulation group (Experimental): Patients in the stimulation group will be stimulated immediately after implantation of the Stimulator (ACTIVA® PC neurostimulator (Model 37601))
  Interventions: Device: ACTIVA® PC neurostimulator (Model 37601)
- Non-stimulation group (Sham Comparator): Patients in the non-stimulation group will not be stimulated for the first three months after implantation of the Stimulator (ACTIVA® PC neurostimulator (Model 37601))
  Interventions: Device: ACTIVA® PC neurostimulator (Model 37601)

INTERVENTIONS:
Device: ACTIVA® PC neurostimulator (Model 37601) — the stimulator in the stimulation group will be turned on after implantation of the device

SUMMARY:
The aim of the study is to prove the efficacy and safety of pallidal DBS in HD patients and to show superiority of DBS on motor function in the stimulation group compared to stimulation-off group

DETAILED DESCRIPTION:
In this study the efficacy and safety of pallidal Deep Brain Stimulation (DBS) in HD patients shall be investigated and superiority of DBS on motor function in the stimulation group compared to the stimulation-off group shall be shown. This study is a prospective, randomised, double blind, parallel group, sham-controlled, multi-centre trial. Patients in the stimulation group will be stimulated for three months while the stimulator in the sham-group will be turned off for three months. After three months the primary endpoint will be assessed. Afterwards the stimulator will be turned on in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically symptomatic and genetically confirmed HD (number of CAG repeats ≥ 36)
* Age ≥18 years
* Moderate stage of the disease (UHDRS motor score ≥ 30)
* Chorea despite best medical treatment (UHDRS chorea subscore ≥ 10)
* Mattis Dementia Rating Scale ≥ 120 (or > 80% of items testable independently from motor impairment)
* Patient has stable medication prior six weeks before inclusion
* Signed informed consent

Exclusion Criteria:

* Juvenile HD (Westphal variant) or predominant bradykinesia
* Postural instability with UHDRS retropulsion score > 2
* Severe comorbidity compromising operability and/or life expectancy and/or quality of life during the trial duration (e.g. cancer with life expectancy < 6 months, NYHA 3 and 4 rising the anaesthetic risk according to the anaesthesiologist)
* Acute suicidality
* Acute psychosis (symptoms within previous 6 months)
* Participation in any interventional clinical trial within 2 months before screening
* Cortical atrophy grade 3
* Patients with risk of coagulopathies and/or increased risk of haemorrhage
* Patients with an implanted pacemaker or defibrillator
* Pregnancy
* lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
UHDRS-TMS difference | 12 weeks postoperatively compared to baseline
  Difference between the groups in the UHDRS total motor score (UHDRS-TMS) at 12 weeks postoperatively compared to baseline.

SECONDARY OUTCOMES:
UHDRS-Chorea difference | 6 months postoperatively compared to baseline
  Difference in the Unified Huntington's Disease Rating Scale (UHDRS) chorea subscore (items 14-20)
UHDRS-bradykinesia difference | 6 months postoperatively compared to baseline
  Difference in the UHDRS bradykinesia subscore (items 22-25 and 27-29)
BFMDRS difference | 6 months postoperatively compared to baseline
  Difference in the Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) motor score
Reilmann Battery differences | 6 months postoperatively compared to baseline
  Difference in the Q-Motor "choreomotography" test (Reilmann Battery)
MDRS difference | 6 months postoperatively compared to baseline
  Difference in the Mattis Dementia Rating Scale (MDRS)
Verbal Fluency Test difference | 6 months postoperatively compared to baseline
  Difference in the Verbal Fluency Test (formal lexical, categorical, category change)
SDMT difference | 6 months postoperatively compared to baseline
  Difference in the Symbol Digit Modalities Test (SDMT)
STROOP Test differences | 6 months postoperatively compared to baseline
  Difference in STROOP word reading, colour naming and colour of the word naming
HADS-SIS difference | 6 months postoperatively compared to baseline
  Difference in the Hospital Anxiety and Depression Scale combined with Snaith Irritability Scale (HADS-SIS)
PBA-s difference | 6 months postoperatively compared to baseline
  Difference in the Problem Behaviours Assessment Short Form (PBA-s)
SF 36 difference | 6 months postoperatively compared to baseline
  Difference in the Short Form (36) Health Survey (SF-36)
CGI difference | 6 months postoperatively compared to baseline
  Difference in the Clinical Global Impression Scale (CGI)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vesper, Prof Dr., Study Chair — Dept. of Functional Neurosurgery and Stereotaxy; Alfons Schnitzler, Prof Dr, Principal Investigator — Dept.of Neurology
Locations (12):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- France (2):
  - CHU Amiens Hôpital nord, Department of neurosurgery and Department of neurology, Amiens
  - Hôpital Roger Salengro, Service de Neurologie et Pathologie du mouvement, Lille
- Germany (7):
  - Charité Campus Virchow Klinikum, Berlin
  - University hospital Heinrich Heine University Düsseldorf, Düsseldorf
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Schleswig-Holstein, Kiel
  - Universität zu Lübeck, Lübeck
  - University hospital Munich LMU, Munich
  - kbo-Isar-Amper-Clinic Taufkirchen, Taufkirchen
- Switzerland (2):
  - Center for Neurology, Bern, Gümlingen
  - Inselspital, Department of Neurology, Bern

IPD SHARING:
Plan to Share IPD: Yes
After the study the data will be provided to the CHDI. The Foundation may use, and make available for use by the Foundation Collaborators, the Study Data for the following purposes: (A) to design and guide future research studies and clinical trials and (B) to support and enable the following scientific discussion and research: (1) to better understand HD or other diseases being studied, (2) that furthers the development of treatments for HD or other diseases or (3) that furthers biomedical research.

REFERENCES:
- [Background] Moro E, Lang AE, Strafella AP, Poon YY, Arango PM, Dagher A, Hutchison WD, Lozano AM. Bilateral globus pallidus stimulation for Huntington's disease. Ann Neurol. 2004 Aug;56(2):290-4. doi: 10.1002/ana.20183. PMID 15293283
- [Background] Groiss SJ WL, Suedmeyer, M, Ploner M, Reck C, Voges J, SturmV, Timmermann L, Schnitzler A. Effect of bilateral pallidal deep brain stimulation in Huntington's disease: A case report. Mov Disord, Volume 21, Issue S15. Tenth International Congress of Parkinson's Disease and Movement Disorders. Kyoto 2006.
- [Background] Fasano A, Cadeddu F, Guidubaldi A, Piano C, Soleti F, Zinzi P, Bentivoglio AR. The long-term effect of tetrabenazine in the management of Huntington disease. Clin Neuropharmacol. 2008 Nov-Dec;31(6):313-8. doi: 10.1097/WNF.0b013e318166da60. PMID 19050408
- [Background] Wojtecki L, Groiss SJ, Ferrea S, Elben S, Hartmann CJ, Dunnett SB, Rosser A, Saft C, Sudmeyer M, Ohmann C, Schnitzler A, Vesper J; Surgical Approaches Working Group of the European Huntington's Disease Network (EHDN). A Prospective Pilot Trial for Pallidal Deep Brain Stimulation in Huntington's Disease. Front Neurol. 2015 Aug 18;6:177. doi: 10.3389/fneur.2015.00177. eCollection 2015. PMID 26347707
- [Background] Wojtecki L, Groiss SJ, Hartmann CJ, Elben S, Omlor S, Schnitzler A, Vesper J. Deep Brain Stimulation in Huntington's Disease-Preliminary Evidence on Pathophysiology, Efficacy and Safety. Brain Sci. 2016 Aug 30;6(3):38. doi: 10.3390/brainsci6030038. PMID 27589813
- [Derived] Kinfe T, Del Vecchio A, Nussel M, Zhao Y, Stadlbauer A, Buchfelder M. Deep brain stimulation and stereotactic-assisted brain graft injection targeting fronto-striatal circuits for Huntington's disease: an update. Expert Rev Neurother. 2022 Sep;22(9):781-788. doi: 10.1080/14737175.2022.2091988. Epub 2022 Jun 29. PMID 35766355
- [Derived] Rodrigues FB, Ferreira JJ, Wild EJ. Huntington's Disease Clinical Trials Corner: June 2019. J Huntingtons Dis. 2019;8(3):363-371. doi: 10.3233/JHD-199003. PMID 31381524
- [Derived] Hartmann CJ, Groiss SJ, Vesper J, Schnitzler A, Wojtecki L. Brain stimulation in Huntington's disease. Neurodegener Dis Manag. 2016 Jun;6(3):223-36. doi: 10.2217/nmt-2016-0007. Epub 2016 May 27. PMID 27230813